CLINICAL TRIAL: NCT00423982
Title: Rifampin Combination Therapy Versus Monotherapy in Early Staphylococcal Infections After Total Hip and Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1603
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Prosthesis-related Infections; Staphylococcal Infections
MeSH Terms: conditions — Prosthesis-Related Infections; Staphylococcal Infections | interventions — Rifampin; Cloxacillin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifampicin-combination therapy (Active Comparator): Cloxacillin or vancomycin in combination with Rifampicin. Treatment of early staphylococcal prosthetic joint infections in addition to debridement and retention of the prosthesis.
  Interventions: Drug: Rifampin-combination therapy
- Monotherapy (Active Comparator): Cloxacillin or vancomycin in the treatment of early staphylococcal prosthetic joint infections in addition to debridement and retention of the prosthesis.
  Interventions: Drug: Monotherapy

INTERVENTIONS:
Drug: Rifampin-combination therapy — Rifampin 300 mg x 3 po and cloxacillin 2 g x 4 iv for two weeks. Then rifampin 300 mg x 3 po and cloxacillin 1 g x 4 po for 4 weeks. In case of methicillin resistance, rifampin 300 mg x 3 po and vancomycin 1 g x 2 iv for 6 weeks.
  Other Names: Antimicrobial therapy in prosthetic joint infection.; Rifampicin and prosthetic joint infection.
  Arms: Rifampicin-combination therapy
Drug: Monotherapy — Cloxacillin 2 g x 4 iv for two weeks, then cloxacillin 1 g x 4 po for 4 weeks. In case of methicillin resistance, vancomycin 1 g x 2 iv for 6 weeks.
  Other Names: Antimicrobial therapy in prosthetic joint infections.; Cloxacillin.; Vancomycin.
  Arms: Monotherapy

SUMMARY:
The number of patients requiring joint replacement is increasing due to its success in restoring function and pain relief, and the growing population of the elderly. One of the most serious complications of arthroplasty is joint prosthesis infection. Due to the absence of prospective, randomized, controlled studies, there is no consensus concerning diagnosis and treatment of prosthetic joint infections. The main objective of this trial is to evaluate the clinical efficacy of rifampin combination therapy versus monotherapy using cloxacillin or vancomycin in early staphylococcal infections after total hip and knee arthroplasty.

DETAILED DESCRIPTION:
The study is a controlled randomized multicentre trial with 8 participating centres in Norway. We will include patients with the diagnosis of early infections (within 4 weeks post operatively)after hip or knee replacement. Patients with clinical signs of infection are scheduled for a standardized soft tissue revision. Diagnosis of staphylococci must be established by arthrocentesis or at surgical revision, and must grow in at least 2/8 cultures.The patients will randomly be assigned to antimicrobial therapy with or without rifampin by a randomization programme. Antibiotics will be given for 6 weeks. Two years follow-up. The study end points are final follow-up visit after two years or relapse of infection.

ELIGIBILITY:
Inclusion Criteria:

* Prosthetic joint infections category 2 or 3 (early post.op infections within 4 weeks).
* Diagnosis of staphylococci.
* Clinically and radiographically stable implants kept in place after revision.

Exclusion Criteria:

* Infection with other microorganisms than staphylococci.
* Less than 2 years of expected survival.
* Predictable inability to comply with the treatment and/or follow-up visits.
* Contraindication to the use of study medication including acute or chronic liver disease.
* Lack of written consent.
* Fertile women.
* Patients taking less than 80% of the study medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-04; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cure defined as lack of clinical, biochemistry or radiological signs of infection at two years follow-up. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Finnur Snorrason, M.D, Ph.D, Study Director — Ullevaal University Hospital
Locations (8):
- Norway (8):
  - Buskerud Central Hospital, Drammen
  - Elverum Hospital, Elverum
  - Martina Hansen Hospital, Gjettum
  - Ringerike Hospital, Hønefoss
  - Lillehammer Hospital, Lillehammer
  - Oslo University Hospital, Ulleval, Oslo
  - Asker and Bærum Hospital, Rud
  - St.Olav Hospital, Trondheim

REFERENCES:
- [Derived] Karlsen OE, Borgen P, Bragnes B, Figved W, Grogaard B, Rydinge J, Sandberg L, Snorrason F, Wangen H, Witsoe E, Westberg M. Rifampin combination therapy in staphylococcal prosthetic joint infections: a randomized controlled trial. J Orthop Surg Res. 2020 Aug 28;15(1):365. doi: 10.1186/s13018-020-01877-2. PMID 32859235